CLINICAL TRIAL: NCT05834582
Title: Neoadjuvant Fluzoparib Combined With Chemotherapy in Germline BRCA-mutated Three-negative Breast Cancer Breast Cancer: an Open, Multicenter, Cohort Trial
Brief Title: Neoadjuvant Fluzoparib in Germline BRCA-mutated Three-negative Breast Cancer Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Liu Xiaoan, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-050
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: TNBC - Triple-Negative Breast Cancer
Keywords: three-negative Breast Cancer with germline BRCA-mutated
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — EC regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort1: Epirubicin+Cyclophosphamide (Experimental): 2 cycles of EC (Epirubicin+Cyclophosphamide) induced chemotherapy, if tumor response is CR or PR: Epirubicin+Cyclophosphamide for 2 cycles Fluzoparib+Paclitaxel for 2 cycles
  Interventions: Drug: Fluzoparib+Paclitaxel; Drug: Epirubicin+Cyclophosphamide
- Cohort2: Fluzoparib+Paclitaxel (Experimental): 2 cycles of EC (Epirubicin+Cyclophosphamide) induced chemotherapy, if tumor response is SD: Fluzoparib+Paclitaxel for 4 cycles
  Interventions: Drug: Fluzoparib+Paclitaxel; Drug: Epirubicin+Cyclophosphamide

INTERVENTIONS:
Drug: Fluzoparib+Paclitaxel — Fluzoparib+Paclitaxel for 4 cycles if tumor response is SD after 2 cycles of EC induced chemotherapy
Drug: Epirubicin+Cyclophosphamide — Epirubicin+Cyclophosphamide

SUMMARY:
Although many PARP inhibitors did not improve pCR in neoadjuvant studies, it is not an unchallenged conclusion that TNBC does not benefit from use of PARP inhibitors in neoadjuvant therapy.This study is an open-label, two-cohort, multicenter trial. 60 patients with germline BRCA-mutated three-negative early breast cancer are planned to be enrolled and treated with fluzoparib combined with chemotherapy according to tumor response after EC (epirubicin and cyclophosphamide) for 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 18 and ≤ 70 years of age with treatment-naïve breast cancer
2. Histopathologically confirmed early or locally advanced three-negative invasive breast cancer as defined by the ASCO/CAP guidelines while meeting the following conditions:

   HER2 negative: IHC 0/1 + or IHC2 + but ISH negative; ER and/or PR negative (not eligible for endocrine therapy): IHC nuclear staining ≤ 1%
3. Tumor stage: II-III: Primary tumor size: ≥ 2cm
4. ECOG score 0 ~ 1;
5. Centrally confirmed BRCA1 or BRCA2 germline mutation;
6. Eligible level of organ function

Exclusion Criteria:

1. Patients with metastatic breast cancer or bilateral breast cancer or inflammatory breast cancer;
2. Participated in other drug trials or received any anti-tumor therapy within 4 weeks before enrollment, including endocrine therapy, immunotherapy, biological therapy or tumor embolization;
3. Previously received PARPi therapy;
4. History of another primary malignancy;
5. Confirmed history of heart failure or systolic dysfunction (LVEF < 50%); high risk uncontrolled cardiac arrhythmias, such as atrial tachycardia;
6. Female patients who are pregnant or lactating;
7. History of allergy to drugs in this study；

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-08 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
tpCR（ypT0/is ypN0） | 6 months from the patients enrolled
  pCR is defined as the absence of invasive residual disease in the breast and in the axillary lymph nodes (ypT0/is ypN0).

SECONDARY OUTCOMES:
Event-free Survival (EFS) as assessed by Investigator | Up to approximately 3 years
  EFS is defined as the time from enrollment to disease progression or death due to any cause
AEs and SAEs | From enrollment to the surgery (approximately 6 months)
  adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoan Liu, Professor, Principal Investigator — Jiangsu Province Hospital/ The First Affiliated Hospital of Nanjing Medical University
Locations (1):
- JiangSu Province Hospital/ The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No